CLINICAL TRIAL: NCT06985784
Title: Enhancing Patient Well-Being: Feasibility of Virtual Reality in Head and Neck Cancer Patients to Improve Depressive Symptomatology, Anxiety and Pain
Brief Title: Virtual Reality Interventions for the Improvement of Depression, Anxiety and Pain in Patients With Head and Neck Cancer and Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24530; NCI-2025-03568 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24530 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (3D mindfulness VR headset) (Experimental): Participants receive 3D mindfulness VR headset consisting of 6 resilience skills training sessions over 30 minutes TIW for 6-7 weeks then weekly for 4 weeks. Participants also wear a Fitbit activity tracker to monitor heart rate, sleep and activity throughout the study.
  Interventions: Other: Interview; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Virtual Technology Intervention
- Arm B (2D non-immersive VR headset) (Active Comparator): Participants receive 2D non-immersive VR headset consisting of 2 scenarios - walk in the nature and beach TIW for 6-7 weeks then weekly for 4 weeks. Participants also wear a Fitbit activity tracker to monitor heart rate, sleep and activity throughout the study.
  Interventions: Other: Interview; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Virtual Technology Intervention

INTERVENTIONS:
Other: Interview — Ancillary studies
Other: Medical Device Usage and Evaluation — Wear a Fitbit
Other: Questionnaire Administration — Ancillary studies
Other: Virtual Technology Intervention — Receive 3D mindfulness VR headset
  Other Names: Virtual Reality Intervention; Virtual Technology
  Arms: Arm A (3D mindfulness VR headset)
Other: Virtual Technology Intervention — Receive 2D non-immersive VR headset
  Other Names: Virtual Reality Intervention; Virtual Technology
  Arms: Arm B (2D non-immersive VR headset)

SUMMARY:
This clinical trial tests how well a three-dimensional (3D) mindfulness virtual reality (VR) versus (vs) two-dimensional (2D) non-immersive interventions works in improving depression, anxiety, pain, and/or stress in patients with head and neck cancer (HNC) undergoing radiation or chemoradiation (C/RT), and their caregivers. HNC patients undergoing C/RT can experience higher levels of depression, anxiety, distress and pain that negatively impact their quality of life. VR allows for a realistic experience and works as an effective distraction tool from the state of pain or anxiety without use of drugs and with minimal associated risk to patients. VR has been shown to help reduce symptoms of depression, anxiety and pain in non-cancer patients, however there is limited evidence of how well VR use works in cancer patients, especially in patients undergoing C/RT for HNC. Caregivers of these patients also experience high levels of anxiety and distress. Using VR interventions may improve depression, anxiety, pain and/or stress in patients with HNC undergoing C/RT and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Feasibility and acceptability of 3D mindfulness VR- vs 2D in HNC patients undergoing C/RT.

SECONDARY OBJECTIVES:

I. Assess patient- and caregiver-preference for 3D VR and non-immersive interventions.

II. Preliminary efficacy in reduction in depressive symptoms, anxiety and pain.

OUTLINE: Participants are assigned to 1 of 2 arms.

ARM A: Participants receive 3D mindfulness VR headset consisting of 6 resilience skills training sessions over 30 minutes three times a week (TIW) for 6-7 weeks then weekly for 4 weeks. Participants also wear a Fitbit activity tracker to monitor heart rate, sleep and activity throughout the study.

ARM B: Participants receive 2D non-immersive VR headset consisting of 2 scenarios - walk in the nature and beach TIW for 6-7 weeks then weekly for 4 weeks. Participants also wear a Fitbit activity tracker to monitor heart rate, sleep and activity throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* PATIENTS: ≥ 18 years
* PATIENTS: Self-reported normal or corrected to normal vision and hearing
* PATIENTS: Ambulatory (permitted to use walking aids such as cane or crutch)
* PATIENTS: Ability to read and understand English for questionnaires
* PATIENTS: Scheduled to undergo C/RT for their HNC
* CAREGIVERS: Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* CAREGIVERS: ≥ 18 years
* CAREGIVERS: Self-reported normal or corrected to normal vision and hearing
* CAREGIVERS: Ability to read and understand English for questionnaires
* CAREGIVERS: A care giver identified by the patient and defined as a person who knows the patient well and is involved in the patient's medical care

Exclusion Criteria:

* PATIENTS: An employee who is under the direct/ indirect supervision of the principal investigator (PI)/ a co-investigator/ the study manager
* PATIENTS: A direct study team member
* PATIENTS: Inability to complete the surveys
* PATIENTS: Serious mental illness
* PATIENTS: Previous head and neck cancer treatment
* PATIENTS: History of any psychiatric disease treatment with anti-depressants, substance abuse, post-traumatic stress disorder (PTSD), chronic pain (> 3 months)
* PATIENTS: Cancer in or around the eyes or ears; visual, hearing or cognitive impairment
* CAREGIVERS: An employee who is under the direct/ indirect supervision of the PI/ a co-investigator/ the study manager
* CAREGIVERS: A direct study team member
* CAREGIVERS: Inability to complete the surveys
* CAREGIVERS: Serious mental illness
* CAREGIVERS: History of any psychiatric disease treatment with anti-depressants, substance abuse, PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-11-09 (Estimated); Study Completion 2027-11-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate (Feasibility) | Up to 11 weeks
  Will be considered feasible if ≥ 50% of patients agree to participate. Will be assessed using summary statistics.
Retention rate (Feasibility) | Up to 11 weeks
  Will be considered feasible if ≥ 70% of patients are retained. Will be assessed using summary statistics.
Adherence to three-dimensional (3D) mindfulness virtual reality (VR) intervention (Feasibility) | Up to 11 weeks
  Will be considered feasible if ≥ 50% of patients use the 3D mindfulness VR intervention. Will be assessed using summary statistics.
Completion of electronic patient reported outcomes (ePRO) (Feasibility) | Up to 11 weeks
  Will be considered feasible if ≥ 70% ePRO assessments are completed. Will be assessed using summary statistics.
Acceptability of 3D mindfulness VR intervention | Up to 11 weeks
  Will be considered acceptable if ≥ 50% patients have greater than neutral satisfaction at the end of the study period. Will be assessed using summary statistics.

SECONDARY OUTCOMES:
Preferences for VR based interventions | Up to 30 days after treatment completion
  Will be assessed by interviews to obtain feedback. Descriptive statistics to summarize satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Krupal Patel, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States